CLINICAL TRIAL: NCT06986941
Title: The Effects of Ballet-Based Exercise Training on Respiratory Functions, Balance, Cognitive Functions, Peripheral Muscle Strength, Functional Capacity and Quality of Life in Patients With Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Selva Otsay, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SelvaPhD2025-001
Record Dates: First submitted 2025-05-04; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease (PD)
Keywords: Ballet-based Dance Therapy; Respiratory Function; Balance; Cognitive Function; Quality of Life
MeSH Terms: conditions — Respiratory Aspiration | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ballet-Based Dance Therapy (Experimental): Participants in this arm will engage in an 8-week ballet-based dance therapy program, specifically designed to enhance functional capacity, balance, peripheral muscle strength, cognitive function, and overall quality of life. The program will be conducted twice a week, with each session lasting approximately 60 minutes. The dance exercises will be tailored to meet the needs of individuals with Parkinson's disease, focusing on improving motor skills, flexibility, and coordination. The primary goal is to assess the impact of ballet-based exercises on various parameters such as respiratory function, balance, and muscle strength.
  Interventions: Behavioral: Ballet-Based Dance Therapy
- Standard Care with Exercise Counseling (Active Comparator): Participants in this arm will continue with their standard medical treatment for Parkinson's disease, including pharmacological management and routine care. Additionally, they will receive a one-time exercise counseling session delivered by a physiotherapist and an informational brochure that includes recommendations for general, unsupervised home-based exercises suitable for Parkinson's patients. No structured or supervised exercise sessions will be provided.
  Interventions: Other: Standard Care with Exercise Counseling

INTERVENTIONS:
Behavioral: Ballet-Based Dance Therapy — An 8-week ballet-based dance therapy program designed to improve balance, flexibility, peripheral muscle strength, cognitive functions, and overall functional capacity in Parkinson's disease patients. The therapy will be conducted twice a week, with each session lasting approximately 60 minutes. The exercises will be adapted to the participants' physical abilities and will focus on enhancing motor coordination, strength, and stability through ballet-inspired movements.
  Arms: Ballet-Based Dance Therapy
Other: Standard Care with Exercise Counseling — Participants in the control group will receive standard care for Parkinson's disease, including pharmacological management and routine clinical follow-up. Additionally, they will receive a one-time exercise counseling session and an informational brochure outlining general home-based exercises appropriate for individuals with Parkinson's disease. No supervised or structured exercise sessions will be conducted.
  Arms: Standard Care with Exercise Counseling

SUMMARY:
This study investigates the impact of an 8-week ballet-based dance therapy on people with Parkinson's disease. It aims to assess the effect of ballet on motor and non-motor symptoms, such as balance, cognitive function, functional capacity, and quality of life. The study will provide insights into the potential of ballet therapy as an effective, non-pharmacological treatment for Parkinson's disease.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the effects of an 8-week ballet-based dance therapy on individuals with Parkinson's disease. The intervention will target motor and non-motor symptoms, including functional capacity, balance, cognitive function, and quality of life. Participants will be randomly assigned to either the intervention group or a control group. The intervention group will engage in structured ballet classes, while the control group will receive standard care. Assessments will include measures of respiratory function, body composition, muscle strength, and balance, with evaluations conducted before and after the intervention. The goal is to assess the feasibility and effectiveness of ballet as a therapeutic approach to improve both physical and mental well-being in people with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Diagnosed with Parkinson's disease.
* Modified Hoehn and Yahr stages I to III.
* Willingness to participate and provide informed consent.

Exclusion Criteria:

* Joint deformities or severe movement limitations that prevent participation in dance exercises.
* Mental retardation (severe cognitive impairment).
* Major surgery within the past 6 months.
* Presence of uncontrolled cardiovascular, pulmonary, or oncological diseases.
* Diagnosed visual or auditory impairments affecting balance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity | At baseline and at week 9 (after 8 weeks of intervention)
  Functional capacity will be assessed using the Six-Minute Walk Test (6MWT) according to American Thoracic Society (ATS) guidelines. The total distance walked will be recorded.
Forced Expiratory Volume in 1 Second (FEV₁) | At baseline and at week 9 (after 8 weeks of intervention)
  FEV₁ will be assessed using spirometry and reported in liters (L). FEV1 will be measured according to the guidelines of the American Thoracic Society (ATS) and the European Respiratory Society (ERS).
Forced Vital Capacity (FVC) | At baseline and at week 9 (after 8 weeks of intervention)
  FVC will be assessed using spirometry and reported in liters (L). FVC will be measured according to the guidelines of the American Thoracic Society (ATS) and the European Respiratory Society (ERS).
Tiffeneau Index (FEV₁/FVC Ratio) | At baseline and at week 9 (after 8 weeks of intervention)
  The ratio of FEV₁ to FVC will be calculated using spirometry and reported as a percentage (%).
Peak Expiratory Flow (PEF) | At baseline and at week 9 (after 8 weeks of intervention)
  PEF will be assessed using spirometry and reported in liters per minute (L/min). PEF will be measured according to the guidelines of the American Thoracic Society (ATS) and the European Respiratory Society (ERS).
Forced Expiratory Flow 25-75% (FEF₂₅-₇₅%) | At baseline and at week 9 (after 8 weeks of intervention)
  FEF₂₅-₇₅% will be assessed using spirometry and reported in liters per second (L/s). FEF₂₅-₇₅%will be measured according to the guidelines of the American Thoracic Society (ATS) and the European Respiratory Society (ERS).

SECONDARY OUTCOMES:
Respiratory Muscle Strength | At baseline and at week 9 (after 8 weeks of intervention)
  Respiratory muscle strength will be assessed by measuring maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) using a digital mouth pressure device, in accordance with established respiratory assessment guidelines.
Balance | At baseline and at week 9 (after 8 weeks of intervention)
  Balance performance will be assessed using the Biodex Balance System. Stability indices will be calculated to evaluate postural control and balance.
Cognitive Function | At baseline and at week 9 (after 8 weeks of intervention)
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA). The MoCA is a 30-point scale ranging from 0 to 30, where higher scores indicate better cognitive performance.
Peripheral Muscle Strength | At baseline and at week 9 (after 8 weeks of intervention)
  Peripheral muscle strength will be assessed using a hand-held dynamometer for major lower extremity muscle groups.
Change in Quality of Life | At baseline and at week 9 (after 8 weeks of intervention)
  Quality of life will be assessed using the Parkinson's Disease Questionnaire-39 (PDQ-39). The total score ranges from 0 to 100, with higher scores indicating worse quality of life.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Podlewska AM, Batzu L, Soukup T, Sevdalis N, Bakolis I, Derbyshire-Fox F, Hartley A, Healey A, Woods A, Crane N, Pariante C, Ray Chaudhuri K. The PD-Ballet study: study protocol for a randomised controlled single-blind hybrid type 2 clinical trial evaluating the effects of ballet dancing on motor and non-motor symptoms in Parkinson's disease. BMC Complement Med Ther. 2024 Jan 17;24(1):41. doi: 10.1186/s12906-023-04296-y. PMID 38233784
- [Background] McGill A, Houston S, Lee RYW. Effects of a ballet-based dance intervention on gait variability and balance confidence of people with Parkinson's. Arts Health. 2019 Jun;11(2):133-146. doi: 10.1080/17533015.2018.1443947. Epub 2018 Mar 6. PMID 31038440